CLINICAL TRIAL: NCT05818527
Title: Effectiveness of Low Frequency Vibration on the Rate of Canine Retraction : A Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Low Frequency Vibration on the Rate of Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: mohamed abdelmotaleb (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, mohamed abdelmotaleb, principle investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: tooth acceleration
Record Dates: First submitted 2023-02-28; First posted 2023-04-19 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- vibrating device arm (Experimental): the patients will use vibrating device 20 mins per day
  Interventions: Device: Acceledent vibrating device
- control group (No Intervention): control group using no devices

INTERVENTIONS:
Device: Acceledent vibrating device — used to accelerated the movement of teeth during orthodontic treatment
  Arms: vibrating device arm

SUMMARY:
The goal of this Randomized controlled clinical trial is To investigate the effectiveness of AcceleDent Aura vibrating device on rate of canine retraction in orthodontic treatment.. The main question[s] it aims to answer are:

• 1st question In Patients with class II requiring canine retraction it possible to accelerate canine retraction safely using AcceleDent? 2nd question: is accelerating teeth movement effect root condition ? the study will be done on Orthodontic patients with class II requiring canine retraction Excluding Any dental or medical disease affecting tooth movement.

DETAILED DESCRIPTION:
Introduction:

orthodontic tooth movement(OTM) is a process of mechanically-induced bone modeling where new bone is formed on the tension side and resorbation on the compression side of the periodontal ligament.

One of negative points of orthodontic treatment is long time treatment (24 month ).

Accelerating the speed of orthodontic tooth movement should contribute to the shortening of the treatment period Many approaches was used such as approaches with low-energy laser irradiation and magnetic fields as well as pharmacological approaches with the injection of prostaglandin E2 (PGE2) and However, many side effects, such as local pain, severe root resorption and drug-induced side effects have been reported.

A new device called AcceleDent(OrthoAccel technologies,Inc, USA) has been introduced to the market and aims to achieve an increased rate of tooth movement by enhancing bone remodelling using pulsating forces. Invented by Dr. Jeremy Mao, it is intended to be used by a patient in conjunction with fixed orthodontic appliances or removable sequential aligner treatment for 20 mins per day. It vibrates at a frequency of 30Hz and has force amplitude of 20 grams.

It was found in kau et al ( split mouth study trial) in that the total rate of movement for the mandibular crowding was 2.1 mm per month and for the maxillary arch was 3.0 mm per month, which apparently is faster than the traditional finding as of about 1.0 mm per month . The patient compliance was 67% with good patient perception. It was thus concluded that the AcceleDent device is a useful adjunct to orthodontic treatment.

The prolonged time of orthodontic treatment especially during extraction cases requiring canine retraction become a major challenge which have not been solved in clinical orthodontic, solving this challenge using AcceleDent will decrease the treatment time of canine retraction thus improve the quality of orthodontic care and improve patient compliance.

Our aim is evaluating the efficiency of device in accelerating tooth movement and shorting time of canine retraction.

Research Hypothesis:

The vibratory stimulation using AcceleDent can accelerate canine retraction, Animal studies have shown that the application of cyclical forces in conjunction with an orthodontic force could increase the rate of orthodontic tooth movement by enhancing bone remodeling activity .

PICOS P- Patients with class II requiring canine retraction I- accelerating canine retraction using AcceleDent C Patients with class II requiring canine retraction using nickel titanium closed spring without AcceleDent O 1ry rate of canine retraction in mm per month. 2ry assist inflammatory root resorption using root resorption index.

Trial design:

Randomized controlled trial

Study setting:

The study will be performed in the outpatient clinic of the Orthodontic Department at the Faculty of Oral and Dental Medicine, Cairo University

Eligibility Criteria:

* Subjects will be on the following inclusion criteria:

  1. Complete permanent dentition
  2. Class II malocclusion that needs first premolar extraction and canine retraction
  3. Subjects with clinically acceptable oral hygiene ( probing depth not exceed 3mm)
* Subjects will be excluded from the study if the following conditions existed:

  1. Any medical could impact study results during the expected length of the study.
  2. Subject was currently using any investigational drug that influence tooth movement (Bisphosphonates, Acetaminophen)15 or any other investigational device.
  3. Subject had plans to relocate or move within 6 months of enrollment.

Intervention:

1. All the patients who will met inclusion and exclusion criteria will be randomly assigned into 2 groups; control and experimental group.
2. For each patient, MBT prescription preadjusted brackets with 0.022*0.025 inch slot (3m Gemini metal brackets, 3m Unitek Corporation, Monrovia, A, USA) will be bonded on the teeth after the first premolars extraction by (T.I)
3. For anchorage preparation, TADs will be used(it will be placed between mesil upper first On the sides requiring anchorage supplementation,1.6-mm TADs (American Orthodontic,US) were placed under local anesthesia, usually at the junction of the attached gingivae with the reflected mucosa and mesially to the maxillary molars. The TADs will be placed before any retraction force placed on the canines16 by (T.I).
4. The canine retraction will be done using Ni-Ti closing spring (3m Unitek Corporation, Monrovia, A, USA),150 gms of force will be used17.
5. The experimental group will be instructed for using AcceleDent from the time of starting canine retraction for 20 mins/day.
6. An alginate impression for the upper arch will be taken monthly. The plaster models will be collected (T0-T4) were digitized using desktop scanner (3Shape R500, 3shape, Copenhagen, Denmark) The canine retraction was assessed using two methods; the incremental rate of canine retraction and the total distance travelled by the canine. Using the 3Shape OrthoAnalyzer software‡ the four consecutive models (T1-T4) were superimposed9 on the base model (T0) using three points registration upon the third rugae area . Colour-mapped superimposition was used to verify the accuracy of the superimposition. The difference in the position of the canine cusp tip was used to calculate the incremental rate of canine retraction (Figure 3). For intra- and inter-rater reliability, measurements of the digital models will done by the same operator (NA) twice, 2 weeks apart and repeated by another operator (MA).

.Measurements of the total distance of canine retraction, the canine tipping, torque and rotation were analysed by measuring the angles between the long axis lines for the canines and the three reference planes were measured to detect tipping and torque movements. Also, the angle between the horizontal line of the first molar and the sagittal plane to detect canine rotation.

For assessment of root resorption, the axial guided navigation method explained by Castro et al10 and Schwartz et al11 was used. Using the software In-vivo , version 5.3(Anatomage, Inc., Santa Clara, CA 95054, USA). the pre- & post-retraction CBCTs obtained for each patient were used to evaluate the effect of AcceleDent on root resorption, the linear length between the root apex and cusps tip was measured.

The evaluation was carried by two blinded examiners. In order to fully visualize the root, the CBCT image was re-oriented on each root so that the cross-section would pass through the long axis of each canine .

The degree of pain was measured by Visual Analog Score (VAS), these charts were filled by the patients for the following week after beginning of canine retraction at time intervals (0, 24 hours , 48 hours, 72 hours and 7 days ) and were gathered at the end of the week. The pain VAS was in the format of a chart that contained a series of 10-cm horizontal scales on which the patient marked the degree of pain (0 to 10, where 0 refer to no pain and 10 refer to sever pain) at the indicated time periods.

Criteria for discontinuing or modifying the allocated intervention:

Patient who had active peridontitis or loss of any of permanent tooth (except third molar) or dental trauma or failure of bonding on maxillary canine during experiment will have to stop the trial.

Adherence:

The patients will be asked to attend regular follow up visits and their adherence to the appointments will be regularly monitored. The patient adherence to intervention instruction ( to use the appliance 20 mins/day) will be monitored by asking the patient and writing every day on chart how long he/she used it?

Outcomes:

Out come Measurement

1. ry Canine retraction mm per month
2. ry Root resorption R.R index

Participant timeline:

Visit Treatment Models CBCT

1. Initial records Yes Yes
2. Brackets and wire placement after premolar extraction Yes No

T0 Start canine retraction In experimental group start the use of acceledent Yes N o 4 T1 1 month after retraction Yes No 5 T2 2 month after retraction Yes No 6 T3 3 month after retraction Yes No 7 T4 4 month after retraction Yes No 8 T5 5 month after retraction Yes No 9 T6 6 month after retraction Yes Yes

Sample size calculation The aim of the study is to evaluate the efficiency of using vibrating device (AcceleDent) in accelerating canine retraction. Based on previous studies the outcome variable is normally distributed and an expected effect size of approximately 0.8. A total sample size of 52 canines will be sufficient to detect a large effect size (d=0.8) estimated from published paper by Kau et al., with power 80% and 5% significance level. This number has been increased to a total sample size of 64 canines (32 in each of the two groups) to allow for losses of around 25% during follow up.

Sample size was calculated using G*Power program, University of Düsseldorf, Düsseldorf, Germany (Faul, F., et.al.).

Statistical methods:

Data management and Statistical analysis will be done using Statistical Package for Social Sciences, Version 21.0 (SPSS, IBM) for Windows. Canine retraction in mm will be presented as mean and standard deviation (SD) or median and range, as appropriate. Percentages will be calculated for inflammatory root resorption.

Differences between continuous variables will be done by Student's t test or Mann-Whitney U-test variables as appropriate. The differences between percentages will be tested using the Chi square test or Fisher's exact test, as appropriate.

P-value <0.05 will be considered statistically significant. All tests will be two-sided.

Allocation:

Sequence generation:

Patients will be randomly assigned to group A (treatment) or B (control) using computer randomization sequence generation into 1:1 at Random.org

Concealment mechanism:

Using sequentially numbered opaque sealed envelopes after signing the informed consent to be enrolled in the study. According to the number, the patients will be then allocated into one of the groups using a randomization table.

Implementation:

The allocation sequence will be generated by a E.Z (Secretary of the orthodontic department) who is not involved in the study. This will be contacted to implement the allocation Blinding : ( the operator and assessor will blinded )

* The operator will be blinded from both groups, (M.N) will be responsible for giving the patient appliance and the follow up of his adherence to instruction
* Only the patients will not be blinded due the nature of the trial
* The assessor (T.F) will be blinded from both the intervention and also the groups

Data collection method:

CBCT ( Siron CBCT, Sirona Dental Systems Inc, New York, USA) and casts

Plans to promote participants retention and complete follow-up:

Telephone numbers of all patients included in the study will be recorded. All patients will be given reminder phone calls at the time of the predetermined follow up dates.

Data management:

* All data will be entered in the computer at the Orthodontic department.
* Resulted data from CBCT, casts analysis will be organized and stored.
* The patients' data should have sequential numbers that will be revised at each step to avoid any mixing of data between patients

Harms:

The patient will be informed in the consent about the 2ry outcome that will be assessment of root resorption , which has not been yet reported in the literature

Interim Analysis:

No interim analysis is to be performed.

Auditing:

The study supervisors will review the trial. The processes to be reviewed will include participant enrolment, consent, eligibility and allocation to study groups; adherence to trial interventions and policies to protect participants, including reporting of harms.

Research ethics approval:

This protocol will be reviewed, approved and agreed upon by CEBD [Center For Evidence Based Dentistry CU] Cairo University, Egypt, and approved by the Ethics Committee [Research Ethics Committee Cairo University Faculty of Oral and Dental Medicine].

Protocol amendments:

Any modifications to the protocol will be agreed upon by the Orthodontics and Dentofacial Orthopedics department.

Consent The trial will be explained to the patients. The researcher will discuss the interventions and possible harms with patients. The researcher will obtain written consent from the patients' parents willing to participate in the trial.

Confidentiality:

All study-related information will be stored securely at the Orthodontic department. All participant personal information will be of limited access. Access will be limited to the minimum number of individuals. All records that contain names will be stored to secure the blinding of analysis.

Declaration of interests:

No financial conflicts of interests are to be declared. The study is self-funded by the researchers.

Access to data:

The researcher and supervisors will have access to the final data sets. All data sets will be password protected. All the data have to be of no access to others until the study is finished.

Ancillary and post-trial care:

All the patient will complete their treatment at out patient clinic Dissemination policy Trial results will be available and A copy of the thesis will be available at the faculty library.

The authors will publish the trial results in angle orthodontics

Funding:

The trial will be self-funded

ELIGIBILITY:
Inclusion Criteria:

Full permanent dentition. Good general and oral health. Severe crowding or protrusion requiring first premolars extractions

Exclusion Criteria:

* Systemic disease or syndrome.

  * Abnormalities in teeth size and/or shape.
  * Vertical, transverse or antero-posterior skeletal discrepancies.
  * History of previous orthodontic treatment.
  * Anti-inflammatory medication

Ages: 15 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amr R Elbialy, professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalajzic Z, Peluso EB, Utreja A, Dyment N, Nihara J, Xu M, Chen J, Uribe F, Wadhwa S. Effect of cyclical forces on the periodontal ligament and alveolar bone remodeling during orthodontic tooth movement. Angle Orthod. 2014 Mar;84(2):297-303. doi: 10.2319/032213-234.1. Epub 2013 Aug 12. PMID 23937517
- [Background] Miles P, Smith H, Weyant R, Rinchuse DJ. The effects of a vibrational appliance on tooth movement and patient discomfort: a prospective randomised clinical trial. Aust Orthod J. 2012 Nov;28(2):213-8. PMID 23304970

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vibrating Device Arm | Control Group
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Afrocentric female Egyptian patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Vibrating Device Arm | Control Group | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (5.1) | 17 (4.1) | 19 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  Egypt | 16 | 16 | 32
canine retraction in millimeter [Mean (Standard Deviation); unit: millimeters] | 5.38 (1.2) | 5.1 (1.1) | 5.28 (1)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Canine Retraction in mm Per Month
Description: . Retraction of the canine was done using NiTi coil spring delivering a force of 150 gm per side calibrated using digital force gauge, attached between the hook of the canine bracket and the first molar tube on a of 16*2 stainless steel basal archwire. The intervention group subjects were given AcceleDent devices which delivered gentle micropulses (0.25 N at 30 Hz) and were instructed to wear them every day for 20 mins according to the manufacturer instructions. The patient compliance to intervention instructions were monitored by asking the patient and writing every day on chart how long she used it and compare this with the data download from the appliance that recorded their daily usage during the period of space closure.
  Follow-up visits were scheduled every four weeks. At each follow up visit, recalibration of the NiTi retraction spring was done using the same force gauge when necessary to maintain 150 gm force delivery. TADs stability and occlusal interferences during canine
Time Frame: 6 month
Population: 32 female patients requiring extraction of upper first premolar
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Vibrating Device Arm | Control Group
Number analyzed (Participants) | 16 | 16
millimeters | 5.38 (1.2) | 5.1 (1.4)

ADVERSE EVENTS:
Time Frame: 6 month
Description: the root length of canine and molar were assessed using CBCT
Arm/Group | Vibrating Device Arm | Control Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT05818527/Prot_SAP_000.pdf